CLINICAL TRIAL: NCT03123198
Title: Dialectical Behavior Therapy Rutgers University Research Program
Acronym: DBT-RU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Shireen L. Rizvi, PhD, ABPP, Associate Professor of Clinical Psychology, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2019001864
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; suicidal behaviors; dialectical behavior therapy
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dialectical Behavior Therapy (Experimental): All participants receive six months of standard DBT which includes individual therapy, skills training, and as-needed phone consultation.
  Interventions: Behavioral: Dialectical Behavior Therapy

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — DBT is a multimodal comprehensive psychosocial treatment.

SUMMARY:
This protocol establishes a research oriented psychological treatment clinic within the Graduate School of Applied and Professional Psychology (GSAPP), called the Dialectical Behavior Therapy Rutgers University Research Program (DBT-RU). The overall aim of the proposed research is to find ways to improve therapist training in existing treatments for complex and difficult-to-treat problems (e.g., DBT, prolonged exposure), develop new and more effective treatments, and improve understanding of severe psychopathology. Consequently, this proposed research will have four branches: (1) training of research clinicians and evaluation of training methods; (2) training of clinical evaluators for the research studies and evaluation of assessment training methods; (3) assessment of treatment outcome, including assessment of mediators and moderators of change (both clinician and client data); (4) assessment and analyses of psychopathology of subject populations who participate in the DBT-RU.

DETAILED DESCRIPTION:
DBT is an evidence-based and empirically supported treatment for borderline personality disorder (BPD), suicide, and self-injury. DBT is traditionally administered for a minimum of 6 months in an outpatient setting but has been adapted to be used in other treatment settings (e.g., intensive outpatient). DBT consists of multiple key components, including weekly individual therapy, group skills training, and option to engage in out-of-session contact with their provider via telephone to receive coaching on how to use DBT skills to manage real-life issues (e.g., urges to harm self). To date, more than a dozen randomized control trials (RCTs) and quasi-experimental studies have been conducted, and compared to 12 months of treatment as usual (TAU), DBT has been shown to result in significantly greater reduction in frequency and severity of self-injurious behaviors, inpatient hospitalizations, suicidal ideation, and substance abuse (see Panos, Jackson, Hasan, & Panos, 2014 ). This research aims to (1) advance our understanding of underlying mechanisms driving treatment outcomes; (2) isolate the effects of particular components and strategies employed in DBT on various outcomes (e.g., suicide), (3) enhance training and evaluation methods for research clinicians; (4) test to see if benefits in DBT are sustained over a period of time beyond follow-up; and (5) advance our knowledge of how DBT operates in everyday life to reduce day-to-day emotion dysregulation and related target behaviors (e.g., suicidal behavior).

ELIGIBILITY:
Inclusion Criteria:

A. Age 18 years or older. B. Agreement to take part in assessments, videotaping/audiotaping and coding of their sessions by research personnel.

C. Agreement to pay for mental health services at the DBT-RU, and to participate in research assessments as volunteers.

D. Residence within commuting distance of clinic (< 45 minutes) E. Agreement to discontinue other forms of therapy F. Meets criteria for borderline personality disorder (BPD)

Exclusion Criteria:

* A. Clients who need mental health services not available at the DBT-RU, such as treatment for schizophrenia or life-threatening anorexia, or who are currently obtaining optimum professional treatment that should not be ended.

B. Non-English speaking. C. Present DSM-IV diagnosis of Mental Retardation. D. Unable to understand research consent forms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Self-Injurious Thoughts and Behaviors Interview | Past six months
  Interview to assess prevalence rates of suicidal and self-injurious thoughts and behaviors
Structured Clinical Interview for DSM-5 | At baseline, lifetime history is assessed. At 3-months and 6-months, changes to diagnostic status are assessed.
  Interview to assess lifetime and current rates of psychological disorders

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale | Past two weeks
Borderline Symptom List (BSL-23) | Past 1 month
Brief Symptom Inventory (BSI) | Past 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yin Q, Hughes CD, Rizvi SL. Using GIMME to model the emotional context of suicidal ideation based on clinical data: From research to clinical practice. Behav Res Ther. 2023 Dec;171:104427. doi: 10.1016/j.brat.2023.104427. Epub 2023 Nov 10. PMID 37980875
- [Derived] Fitzpatrick S, Bailey K, Rizvi SL. Changes in Emotions Over the Course of Dialectical Behavior Therapy and the Moderating Role of Depression, Anxiety, and Posttraumatic Stress Disorder. Behav Ther. 2020 Nov;51(6):946-957. doi: 10.1016/j.beth.2019.12.009. Epub 2019 Dec 30. PMID 33051036